CLINICAL TRIAL: NCT01010074
Title: Intrinsically Photosensitive Retinal Ganglion Cells in Parkinson's Disease
Brief Title: Retinal Function in Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Bruce I. Gaynes, OD, PharmD, Hines VA Medical Center
Organization: Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Other Study IDs: PD001
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Parkinson's Disease
Keywords: retina, Parkinson's disease, ganglion cell, pupillary
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disorder characterized by muscle rigidity, tremor, a slowing of physical movement (bradykinesia) and, in extreme cases, a loss of physical movement. The primary symptoms are the results of decreased stimulation of the motor cortex arising from the basal ganglia normally caused by the insufficient formation and action of dopamine, which is produced in the dopaminergic neurons of the brain. Secondary symptoms may include high level cognitive dysfunction and subtle language problems. Included in the symptomatology experienced by patients with PD, visual abnormalities are not uncommon. Visual changes among patients with PD appear not only dynamic in nature, but differentially affected based on the course of the disease and, perhaps more importantly, its treatment. Parkinson's disease has significant ramifications not only in observation of irregularities in vision, but how vision interacts with entrainment of the circadian clock. The purpose of this study is to examine the relationship between PD and operation of a unique set of retinal cells known to regulate the circadian clock and sleep-wake cycles in human subjects.

ELIGIBILITY:
Inclusion Criteria: age 18-64 best corrected visual acuity of 20/25 or better in each eye -

Exclusion Criteria: evidence of any form of eye disease, inability to understand and sign informed consent.

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: movement disorders/neurology clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
pupillary threshold | one

CONTACTS AND LOCATIONS:
Locations (1):
- Hines VA Medical Center, Hines, Illinois, United States